CLINICAL TRIAL: NCT07115043
Title: A Phase I/II Open-label Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD6750, a CD8 Guided IL-2 Agent Alone and in Combination With Other Anti-cancer Agents in Participants With Select Advanced or Metastatic Solid Tumors
Brief Title: A Study to Investigate Safety of AZD6750 in Adult Participants With Select Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D7350C00001
Record Dates: First submitted 2025-07-16; First posted 2025-08-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma (Skin); Renal Cell Carcinoma; Merkel Cell Carcinoma; Triple Negative Breast Cancer; Head and Neck Squamous Cell Carcinoma; Gastric Cancer/Gastroesophageal Junction Cancer; High Grade Serous Ovarian Carcinoma
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Squamous Cell; Carcinoma, Renal Cell; Carcinoma, Merkel Cell; Triple Negative Breast Neoplasms; Squamous Cell Carcinoma of Head and Neck; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Module 1 consists of treatment with AZD6750 administered as a single agent to enroll participants with select locally advanced or metastatic solid tumors who have received prior adequate SoC. Select solid tumors include the tumor types known to show activity with ICIs (either as a single agent or in combination with other anti-cancer agents) or include reports potentially showing benefit of IL-2. Module 1 will consist of Part 1A (dose escalation). The combination arm (Module 2) will open on agreement with SRC, and will investigate AZD6750 and rilvegostomig, enrolling participants with Stage IV NSCLC who either received at least one line of therapy in metastatic setting or are treatment naïve in metastatic setting and have a PD-L1 expression ≥ 1%. Module 2 will consist of an escalation arm (Module 2A) and an expansion arm (Module 2B). Dose expansion (Module 2B) may open further to characterize preliminary efficacy of AZD6750 in combination with rilvegostomig.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Module 1 (Experimental): AZD6750 administered intravenously (IV) as a single agent
  Interventions: Drug: AZD6750
- Module 2 (Experimental): AZD6750 given in combination with rilvegostomig (IV)
  Interventions: Drug: AZD6750; Drug: rilvegostomig

INTERVENTIONS:
Drug: AZD6750 — AZD6750- CD8 guided IL-2
Drug: rilvegostomig — Rilvegostomig- PD1-TIGIT bispecific antibody
  Arms: Module 2

SUMMARY:
A Study to Investigate Safety of AZD6750 in Adult Participants With Select Advanced or Metastatic Solid Tumors

DETAILED DESCRIPTION:
A Phase I/II Open-label Dose Escalation and Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD6750, a CD8 Guided IL-2 Agent Alone and in Combination With Other Anti-cancer Agents in Participants with Select Advanced or Metastatic Solid Tumors

ELIGIBILITY:
Inclusion criteria:

* Participant ≥ 18 year
* ECOG PS of 0 to 1
* Provision of 'archival' tumor specimen
* At least one measurable lesion according to RECIST v1.1,
* Minimum life expectancy of 12 weeks
* Adequate and stable cardiac function
* Adequate bone marrow, liver and kidney function
* Body weight ≥ 35 kg
* Capable of giving signed informed consent

Module 1 specific inclusion criteria:

• Participants with locally advanced or metastatic select solid tumors (MM, Squamous cell carcinoma of skin, MCC, NSCLC, Head and neck squamous cell carcinoma, Gastric cancer/gastroesophaegeal junction cancer, RCC, HGSOC, Triple negative breast cancer) who have received adequate SoC

Module 2 specific inclusion criteria:

* Participants with Stage IV NSCLC Dose Escalation/Backfills

  1. Have received at least one prior regimen in metastatic setting (2L+ NSCLC). Participants with actionable tumor alterations should have received targeted therapy if locally available OR
  2. Have not received systemic therapy (1L NSCLC) and have PD-L1 expression ≥ 1%.

     Dose Expansion

  <!-- -->

  1. Have not received systemic therapy (1L NSCLC) and have PD-L1 expression ≥ 1%.

     Exclusion criteria:
* Any evidence of:

Severe or uncontrolled systemic diseases including respiratory, cardiac or tumor-related conditions

* History or planned organ or allogeneic stem cell transplantation.
* Active or prior documented autoimmune or inflammatory disorders, within the past 3 years
* Any prior toxicities that led to permanent discontinuation of prior immunotherapy
* Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anti-cancer therapy
* Brain metastases unless treated, asymptomatic, stable, and not requiring continuous corticosteroids
* Acute untreated or symptomatic malignant spinal cord compression, or a history of leptomeningeal carcinomatosis.
* Active uncontrolled or chronic infection of hepatitis B, hepatitis C
* Prior history of Grade ≥ 3 non-infectious pneumonitis.
* Participant requires chronic immunosuppressive therapy (including steroids > 10 mg prednisone/day or equivalent).
* Receipt of live attenuated vaccine within 30 days.

Module 2 specific exclusion criteria:

* Previous treatment with anti-TIGIT therapy
* 1L NSCLC participants with genetic alteration such as EGFR that has a targeted therapy in 1L as per local SoC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-29 (Actual); Primary Completion 2029-10-02 (Estimated); Study Completion 2029-10-02 (Estimated)

PRIMARY OUTCOMES:
Safety- Part 1A & Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from the informed consent until Day 90 post-last dose.
  To assess the safety and tolerability, characterize the DLTs, and determine the MTD and RP2D(s) of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module
Efficacy- Part 2B only (dose expansion) | Measured every 6 weeks for 48 weeks and every 12 weeks thereafter from first dose until disease progression or death in the absence of disease progression(approximately 2 years)
  To assess the preliminary anti-tumor activity of AZD6750 in combination with other anti-cancer agents.

SECONDARY OUTCOMES:
Pharmacodynamic- Part 1A & Part 2A (dose escalation) and Part B (dose expansion) | Measured with baseline and On-treatment biopsy. On-treatment biopsy is planned during Cycle 2 during Cycle 2 (each cycle is 28 days or 21 days depending on Module/dosing schedule)
  To assess immunomodulatory biomarker PD-L1 at baseline and on treatment as a single agent and in combination with other anti-cancer agents as specified in each respective module
Immunogenicity- Part 1A & 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose. Each cycle is 28 days or 21 days depending on Module/dosing schedule).
  To assess the incidence of anti-drug antibodies (ADA) against AZD6750 in serum and in combination with other anti-cancer agents as specified in each respective module
Efficacy (Part 1A and 2A) | Measured every 6 weeks for 48 weeks and every 12 weeks thereafter thereafter from first dose until disease progression or death in the absence of disease progression (approximately 2 years)
  To assess the preliminary anti-tumor activity of AZD6750 alone and in combination with other anti-cancer agents.
PK Maximum plasma concentration (Cmax)- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the plasma concentration of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 days depending on Module/dosing schedule)
PK Area Under Curve (AUC)- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the Area Under Curve (AUC) of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 days depending on Module/dosing schedule.
PK Time to maximum plasma concentration (tmax)- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the time to maximum plasma concentration of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 days depending on Module/dosing schedule.
PK Clearance- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the clearance of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 days depending on Module/dosing schedule.
PK Half-life- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the PK half-time of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 depending on Module/dosing schedule.
PK Minimum observed concentration (Cmin)- Part 1A and Part 2A (dose escalation) and Part 2B (dose expansion) | Measured from pre-infusion on Cycle 1 up to Day 28 post last dose on predefined intervals
  To assess the minimum observed concentration (Cmin) of AZD6750 as a single agent and in combination with other anti-cancer agents as specified in each respective module. Each cycle is 28 days or 21 days depending on Module/dosing schedule.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Research Site, Grand Rapids, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Fairfax, Virginia
- Research Site, East Melbourne, Australia
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kashiwa

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/